CLINICAL TRIAL: NCT02887066
Title: Observatory on Emergency Care for Acute Coronary Syndrome in Grand Est of France
Acronym: CHEST
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/DAIICHI/CHEST-CHOUIHED/MS
Record Dates: First submitted 2016-08-19; First posted 2016-09-01 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-08

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with thoracic pain and suspicion of ACS

SUMMARY:
The purpose is to build up a data observatory of individuals with thoracic pain evoking acute coronary syndrome (ACS). The aim is the characterization of this population of patients consulting at emergency department, the evaluation of therapeutic strategies with regard to guidelines and the becoming of patients including severe complications and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Resident in Grand Est of France (Lorraine, Champagne Ardenne) under medical care at the emergency room or outside of hospital or in cardiology:
* Outside of hospital: for thoracic or epigastric pain with suspicion of ACS Emergency: for thoracic pain for which the doctor will prescribe troponin or troponin kinetics
* Affiliation to social security

Exclusion Criteria:

* Patient affected by ACS with ST segment elevation
* Patient with traumatic thoracic pain
* Patient with thoracic pain of parietal origin
* Patient with consciousness troubles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in emergency room or under medical care in mobile intensive care units for thoracic pain and suspicion of ACS.
Sampling Method: Non-Probability Sample
Enrollment: 580 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
Mortality | 1 year
Severe complications | 30 days
Severe complications | 1 year
Benefit/risk ratio of treatments | day 0
Benefit/risk ratio of treatments | 30 days
Benefit/risk ratio of treatments | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tahar Chouihed, Principal Investigator — Service SAMU - SMUR - SAU, Hôpital Central, CHRU de Nancy

IPD SHARING:
Plan to Share IPD: No